CLINICAL TRIAL: NCT04232397
Title: A Phase 2 Study of Anlotinib in Subjects With Steroid Depenent/Refractory Chronic Graft Versus Host Disease(cGVHD)
Brief Title: Anlotinib Treatment in Steroid Depenent/Refractory cGVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the efficency is not good enough to enroll more patients
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-Anlo-cGVHD-2019001
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Chronic Graft-versus-host-disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- therapy (Experimental): therapy with 1 arm. Anlotinib 8mg qd po。
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — anlotinib 8mg qd po

SUMMARY:
This is a single center, single arm, prospective, phase II clinical study. The main purpose of this study is to evaluate the efficacy and safety of anlotinib in the treatment of steroid dependent/refractory chronic graft-versus-host disease (cGVHD) after allogeneic peripheral blood stem cell transplantation (allo HSCT).

DETAILED DESCRIPTION:
Anlotinib 8mg qd po for 6months if no progression in 4weeks or reach PR in 3months

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be diagnosed as hematopoiesis disorders and receiving hematopoietic stem cells transplantation.
2. Steroid dependent or refractory classic chronic GVHD disease defined as modified National Institutes of Health criteria(2014) below at any time post-hematopoietic cell transplant(post-HCT)

   1. Dependent disease, defined as, when glucocorticoid (prednisolone doses greater than or equal to(<=) 0.25mg/kg/day or <=0.5mg/kg every other day(prednisolone doses) due to recurrence or progression of cGVHD manifestations, it is considered as steroid-dependent disease if the lowest tapering dose of the second occasion is equal or higher than the lowest tapering dose of the first occasion
   2. Refractory disease, defined as, when cGVHD manifestations progress despite the use of a regime containing glucocorticoid (prednisolone at >=1mg/kg/day for at least 1 week) or persist without improvement despite continued treatment with glucocorticoid (prednisolone at >=0.5mg/kg/day or 1mg/kg every other day) for at least 4 weeks.
3. Participants must be receiving baseline systemic glucocorticoid therpy for cGVHD at study entry. The dose of steroids must be stable for 14 days prior to starting anlotinib.
4. At the time of trial enrollment, participants may be receiving other immunosuppressive therapies in addition to glucocorticoids. Immunosuppressant doses must be stable for 14 days prior to starting anlotinib.
5. Neutrophil≥1.5×109/L，platelet≥50×109/L
6. Karnofsky or Lansky performance status>=60
7. Participants should sign the agreement.

Exclusion Criteria:

1. Known or suspected active acute GVHD.
2. Current treatment with a tyrosine kinase inhibitor, purin analogs or other cancer chemotherapy in the 4weeks prior to starting study drug.
3. Concomitant use of warfarin or other Vitamin K antogonists.
4. Known bleeding disorders or hemophilia.
5. Known history of human immunodeficiency virus or active with hepatitis C. virus or hepatitis B virus.
6. Uncontrolled infections not responsive to antibiotics, antiviral medicines, or antifungal medicine or recent infection requiring systemic treatment .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate as the percentage of participants with response. | 1year
  Overall response rate is defined as the proportion of subjects who achieved complete response CR or partial response PR. Response criteria are based on NIH cGVHD Response assessment.

SECONDARY OUTCOMES:
Duration of Response (DOR) | 1year
  DOR is defined as the duration of time from the date of initial response

CONTACTS AND LOCATIONS:
Overall Officials: xianmin song, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Hematology Department, Shanghai, Shanghai Municipality, China